CLINICAL TRIAL: NCT02184221
Title: The Effectiveness of Deep-brain Magnetic Stimulation in the Treatment of Major Depressive Disorder：a Preliminary Study
Brief Title: Deep-brain Magnetic Stimulation (DMS) in the Treatment of Major Depressive Disorder
Acronym: DTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Gang Wang, MD, Head of Depression Center, Vice-principal of, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMS-2010
Record Dates: First submitted 2014-06-30; First posted 2014-07-09 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Major Depressive Disorder
Keywords: Deep-brain magnetic stimulation; Brain derived neurotropic factor; Effectiveness; Safety
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High frequency stimulation (Experimental): alpha burst, 8~12Hz, run 2 seconds, rest 8 seconds, lasts 20 minutes each time
  Interventions: Device: High frequency stimulation
- Low frequency stimulation (Active Comparator): 0.5Hz, run 0.5 seconds, rest 1.5 seconds, lasts 20 minutes each time
  Interventions: Device: Low frequency stimulation

INTERVENTIONS:
Device: High frequency stimulation — The parameter of DMS: alpha frequency
  Other Names: Alpha frequency stimulation
  Arms: High frequency stimulation
Device: Low frequency stimulation — The parameter of DMS: 0.5Hz
  Other Names: 0.5Hz stimulation
  Arms: Low frequency stimulation

SUMMARY:
Transcranial magnetic stimulation (TMS) is an effective alternative for pharmacotherapy in major depressive disorder, but the effectiveness is not clear due to stimulated region, frequency and intensity of magnet field. Standard TMS techniques only can stimulate superficial cortical areas as the electric field decreases rapidly as a function of tissue depth，while depression is also interconnected with deeper neuronal regions. Deep-brain magnetic stimulation (DSM, or deep TMS, DTMS) allows stimulation of deeper cortical regions. Previous research has demonstrated that alpha frequency (8-13 Hz) EEG activity may have particular relevance to the response to antidepressants, and reduction of alpha frequency (8-13 Hz) could lead to negative symptoms. It has been reported that both alpha frequency and low-field magnetic stimulation could improve depressive symptoms.

The objective of this study is to compare the effectiveness of the two different parameters of DMS in the treatment of major depressive disorder. The changes of brain derived neurotropic factor (BDNF) are also investigated to make a relevant analysis of the improvement of depressive symptoms.

DETAILED DESCRIPTION:
The study is designed as randomized, double-blinded, active-controlled trial in major depressive disorder.

Patients will be male or female, 18 to 60 years of age, right-handed, outpatient or inpatient status, with diagnosis of major depressive episode (single or recurrent) by DSM-IV. The HAMD-17 total score is no less than 18 at enrollment. The patients should be drug free at least 30 days before entering the trial. The eligible patients are randomized to one of the two treatment groups using a 1:1 ratio for the alpha frequency (high frequency) and 0.5Hz (low frequency) groups.

Throughout the course of the study, DMS sessions are administered by trained physicians for 20 minutes at a time, with 5 sessions per week, during 6 consecutive weeks. Raters who are blinded to the treatment arm perform evaluations. The effective outcome is assessed by the HAMD-17 and HAMA every two weeks including randomization. Serum BDNF level are also tested at each visits (Week 0, 2, 4 and 6). The safety in this study will be assessed by adverse event reporting, clinical laboratory measurements and physical examinations.

Primary efficacy measure will be assessed based on the decrease of HAMD-17 from randomization to endpoint (Week 6).

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent.
* Aged from 18 to 60 years old.
* Has a diagnosis of major depressive disorder by DSM-IV criteria.
* HAMD-17 ≥ 18.
* Right-handed.
* Be drug free at least 30 days at randomization.

Exclusion Criteria:

* Current Axis I primary psychiatric diagnosis other than major depressive disorder.
* Organic mental disease, including mental retardation.
* History of clinically significant disease, including any cardiovascular, hepatic, renal, respiratory, hematologic, endocrinologic, or neurologic disease, or clinically significant laboratory abnormality that is not stabilized or is anticipated to require treatment during the study.
* Subjects receiving an investigational agent (including different formulation and generic agents of investigational drug) in the previous 3 months prior to screening.
* Women in pregnancy or lactation, or female of child bearing potential without appropriate birth control measures.
* Has received ECT or MECT within 3 months prior to screening.
* Significant risk of suicidal and/or self-harm behaviors.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Improvement of Depression | From randomization to endpoint(Week 6)
  the Change of 17-item Hamilton Depression Scale (HAMD-17) total score

SECONDARY OUTCOMES:
Improvement of Anxiety | From randomization to endpoint (Week 6)
  the Change of Hamilton Anxiety Scale (HAMA) total score
Remission rate | From randomization to endpoint (Week 6)
  The proportion of subjects at endpoint with HAMD-17≤7
Response rate | From randomization to endpoint (Week 6)
  The proportion of subjects at endpoint with the reduction of HAMD-17 total score>=50%
Safety outcome 1 | From enrollment to endpoint (Week 6)
  The incidence and nature of adverse events
Safety outcome 2 | From randomization to endpoint (Week 6)
  The number of subject withdrawal due to adverse events

OTHER OUTCOMES:
BDNF change | From randomization to endpoint (Week 6)
  Change of serum BDNF level

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, M.D., Ph.D, Principal Investigator — Beijing Anding Hospital, Capital Medical University
Locations (1):
- Beijing Anding Hospital, Beijing, Beijing Municipality, China